CLINICAL TRIAL: NCT01542411
Title: Effectiveness of Aspirin in Compare With Heparin Plus Aspirin in Recurrent Pregnancy Loss Treatment
Status: Completed | Type: Observational
Sponsor: Yazd Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2362
Record Dates: First submitted 2012-02-25; First posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Recurrent Pregnancy Loss

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- recurrent pregnancy loss
- thrombophilia, aspirin
- heparin

SUMMARY:
This study evaluated the effect of anticoagulant treatment on the live-birth rate in women with a history of at least two continuous unexplained miscarriages or thrombophilia. It also compared two methods of treatment with aspirin and aspirin plus heparin.

ELIGIBILITY:
Inclusion Criteria:

* unexplained recurrent miscarriage,
* women had previous venous or arterial thromboembolism or who were heterozygous or homozygous for mutations for FV Leiden G1691A, prothrombin gene G20210A (FII G20210A), and methyltetrahydrofolate reductase C677T (MTHFR C677T)

Exclusion Criteria:

* abnormal karyotypes of both partners,
* uterine and cervical anatomical disorders on pelvic ultrasonography or hysteroscopy,
* abnormal ovaries and abnormal endocrine tests.

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This project evaluated 520 women with unexplained recurrent miscarriage for four years. They had referred to recurrent abortion clinic of Yazd Reproductive sciences institute. Women with unexplained recurrent miscarriage included in this study
Sampling Method: Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2008-04

CONTACTS AND LOCATIONS:
Overall Officials: Tahere Jahaninejad, MSC, Principal Investigator — Yazd Shahid Sadoughi Medical Sciences University and Health Services, Yazd, Iran
Locations (1):
- Research and Clinical Centre for Infertility, Yazd, Yazd Province, Iran